CLINICAL TRIAL: NCT06362122
Title: Anatomo-clinico-biological Profiles in Severe Nasal Polyps
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PREDICTO-POLYP
Record Dates: First submitted 2024-02-05; First posted 2024-04-12 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-05

CONDITIONS: NASAL POLYPS
MeSH Terms: conditions — Nasal Polyps

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with nasal polyps (Experimental)
  Interventions: Other: identification anatomo-clinico-biological profiles

INTERVENTIONS:
Other: identification anatomo-clinico-biological profiles — to determine an anatomo-clinico-biological correlation associating the anatomopathological profile, the clinical characteristics and the cytokine signature

SUMMARY:
Nasal sinus polyposis is a chronic inflammatory pathology of the nasal cavity and sinus cavities that causes bilateral and multifocal polyp development and has a prevalence of 2 to 4% in the general population.

Therapeutic management consists of first-line medical treatment for anti-inflammatory purposes. Local corticosteroid therapy, using nasal sprays, is the background treatment. Surgical management is offered to patients in case of failure of medical treatment. Although effective, surgery does not protect patients from recurrence of symptoms related to regrowth of polyps. Recently, biologics have appeared, which despite its effectiveness, about 20% of patients have a partial or no response to these treatments. There is currently no possibility of determining the probability of response to treatments in patients.

It is therefore essential to determine an anatomo-clinico-biological correlation associating the anatomopathological profile, the clinical characteristics and the cytokine signature in order to best guide the patient's management, including the initiation of biotherapy. Indeed, patients, according to their clinical, biological characteristics and the cytokine signature of their polyps will react differently to different treatments, including surgery and biotherapy. This correlation will serve as a predictor of treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 year-old
* Patient with nasal sinus polyposis resistant to medical treatment and requiring surgical treatment with ethmoidectomy type is considered for the first time
* Having signed the consent form
* Having an health insurance

Exclusion Criteria:

* Current or past biotherapy treatment
* Taking general corticosteroid therapy within 4 weeks of surgery
* Protected person
* Pregnant women or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-05-03 (Estimated); Study Completion 2026-10-03 (Estimated)

PRIMARY OUTCOMES:
Identify anatomical profiles present in nasal sinus polyposis resistant to medical treatment. | 1 day
  Caracterization the profiles of patients by the presence or not of edematous or fibrous component, infiltration and lymphoplasmocytic infiltrates.
Evaluation of symptoms related to nasal sinus polyposis by visual analogue scale | 1 day
  the measurement by the visual analogue scale (ranging from 0 (no) to 10 (very intense)
Evaluation to quality of life by Sino-Nasal Outcome Test | 1 day
  the measurement to quality of life by Sino-Nasal Outcome Test (test SNOT-22: test is a questionnaire that reviews 22 symptoms. Each item quantifies the severity of the symptom from 0 (no problem) to 5 (very severe problem). The maximum score is 110, a high score indicating a significant impact of symptoms).
Identify biological profiles for patients with nasal sinus polyposis | 1 day
  The measurement to cytokine expression of naso-sinus polyps (RNA sequencing analysis)
Evaluation to cytokine concentration in serum for patients with nasal sinus polyposis | 1 day
  The measurement to cytokine concentration in serum (mg/l)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Poitiers, Poitiers, France